CLINICAL TRIAL: NCT04546529
Title: Trans-spinal Magnetic Stimulation (TsMS) in Parkinson's Disease- Related Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, MD, PhD (Head of Pain Division), University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JDLDCA
Record Dates: First submitted 2020-07-05; First posted 2020-09-14 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Musculoskeletal Pain; Parkinson Disease
Keywords: non-motor symptom; Musculoskeletal Pain; Parkinson disease; treatment; Trans-spinal Magnetic Stimulation
MeSH Terms: conditions — Musculoskeletal Pain; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TsMS active (Active Comparator): Patients undergoing real Trans-spinal Magnetic Stimulation (TsMS) for 8 weeks
  Interventions: Device: Trans-spinal Magnetic Stimulation (TsMS)
- TsMS sham (Sham Comparator): Patients undergoing placebo Trans-spinal Magnetic Stimulation (TsMS) for 8 weeks
  Interventions: Device: Sham Trans-spinal Magnetic Stimulation (TsMS)

INTERVENTIONS:
Device: Trans-spinal Magnetic Stimulation (TsMS) — Patients undergoing real TsMS with coil
  Arms: TsMS active
Device: Sham Trans-spinal Magnetic Stimulation (TsMS) — Patients undergoing placebo TsMS with coil
  Arms: TsMS sham

SUMMARY:
Parkinson disease is the second most common neurodegenerative disease. Pain is the frequent non-motor symptom that significantly compromises the quality of life, affecting 80% of patients during the course of the disease. There is currently no evidence-based treatment for PD-related pain in general. Nociceptive pain is the most frequent pain in PD an is frequently musculoskeletal in nature. Epidural spinal cord stimulation is known to provide analgesic effects in several types of pain syndromes. Here we test analgesic effects of a non-invasive trans-spinal magnetic stimulation as an add-on treatment for nociceptive (musculoskeletal) pain directly related to Parkinson disease.

DETAILED DESCRIPTION:
Background: pain is frequent non-motor symptom in Parkinson's disease (PD) that significantly compromises the quality of life, affecting 80% of patients during the course of the disease. Nociceptive pain is the most frequent subtype, mainly musculoskeletal in nature. There is currently no evidence-based treatment for PD-related pain in general. The present study tests the effectiveness and safety of non-invasive trans-spinal magnetic stimulation (TsMS) to treat musculoskeletal pain directly related to PD in a sham-controlled randomized approach.

Patients and Methods: this is a randomized, sham-controlled trial including 40 subjects, aged between 18 and 85 years, with musculoskeletal pain directly related to PD, that will be randomized to receive TsMS active or TsMS sham in a 1:1 ratio. Enrollment will take place at the Pain Center of the University of São Paulo and Movement Disorders Center of the University of São Paulo.

We have decided to perform an interim analysis when 24 patients will be included in the trial in order to assess safety and calculate effect size of the active intervention, after meeting with the research and statistical board. A decision will thereafter be made to, either: 1: halt the study due to futility, 2: continue the study with a new target sample size based on the calculations made with the effect from the n= 24 sample.

Expected results: the study hypothesis is that non-invasive trans-spinal magnetic stimulation is superior to sham and it is safe to use that device in patients with nociceptive (musculoskeletal) pain in PD.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease
* Parkinsson disease related musculoskeletal Pain
* Signed term of informed consent

Exclusion Criteria:

* Pregnant or lacting women
* Predominant neuropathic pain
* The presence of psychiatric disorders such as uncontrolled posttraumatic stress disorder, uncontrolled depression, uncontrolled anxiety disorder and suicidal ideation;
* Who wishes at any time to abandon the study;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Number of responders | base line (moment of inclusion) and the last day of the patient assessment (2x in two months)
  Number of individuals presenting 50% pain intensity reduction (on VNS 0-10 average pain of BPI item 5) in the active vs the sham group at the last (8th week) assessment compared to baseline values.

SECONDARY OUTCOMES:
Change in baseline of Pain | base line (moment of inclusion) and in the last day after the final session of TMS-e (2x in two months)
  Assessing by score derivated of Parkinson's Disease Pain Classification System (PD-PCS). This score range from 0 (minimum) to 90 (maximum), being considered an effective improvement in the patient's pain when the pain decreases at least in 50% from the basal score.
Incidence of Treatment-Emergent Adverse Events | Immediately after the intervention (session of stimulation)
  The safety of trans-spinal magnetic stimulation (TsMS) will be assessed by measuring the number of participants who experience serious events. Each serious adverse event be described in detail
Mood | base line (moment of inclusion) and the last day of the sessions of TMS-e (2x in two months)
  Assess mood by hospital anxiety and depression scale
Quality of life related to pain relief | base line (moment of inclusion) and the last day of the sessions of TMS-e (2x in two months)
  Assess by EuroQol- 5 Dimension
Parkinson's disease motor symptoms | base line (moment of inclusion) and the last day of the sessions of TMS-e (2x in two months)
  Assess by UPDRS part III
Interference in daily activities | base line (moment of inclusion) and the last day of the sessions of TMS-e (2x in two months)
  measured by brief pain inventory
Global impression of change | base line (moment of inclusion) and the last day of the sessions of TMS-e (2x in two months)
  Assess % of very much and much improved

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ciampi, PHD, Study Chair — University of São Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The complete IPD will be shared with other authors who wish to use it in individual patient data (IPD) meta-analysis. Other specific situations will be discussed on a case-by-case basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be available after the estimated study completion time (December/2021) and for five years.
Access Criteria: use in individual patient data (IPD) meta-analysis. Other specific situations will be discussed on a case-by-case basis.

REFERENCES:
- [Derived] Lapa JDDS, da Cunha PHM, Teixeira MJ, Brito Medeiros VM, Fernandes AM, Silva de Morais AD, Graven-Nielsen T, Cury RG, Ciampi de Andrade D. Burst Transspinal Magnetic Stimulation Alleviates Nociceptive Pain in Parkinson Disease-A Pilot Phase II Double-Blind, Randomized Study. Neuromodulation. 2023 Jun;26(4):840-849. doi: 10.1016/j.neurom.2022.10.043. Epub 2022 Nov 18. PMID 36411151